CLINICAL TRIAL: NCT06595914
Title: Improving In-hospital and Post-discharge Patient Education for Mild Traumatic Brain Injury
Acronym: EDucate
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency); Ohio State University (Other)
Responsible Party: Principal Investigator, Lindsay Nelson, Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: PRO00051478; HT9425-24-1-0376 (Other Grant/Funding Number: U.S. Army Medical Research Acquisition Activity)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Concussion, Mild; Traumatic Brain Injury
Keywords: Education; Systems of care; Emergency department; Implementation science
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic; Emergencies

STUDY DESIGN:
Intervention Model Description: The study will enroll and follow emergency department clinicians and their patients. Clinicians will be the focus of the intervention.
Who Masked: Participant
Masking Description: Because the intervention disseminates clinical implementation strategies to clinicians, clinicians will not be masked. Patient participants will be masked to whether their outcomes are being collected pre- versus post-clinician intervention. Patient participants will not be masked with regard to having received the mHealth tool for post-discharge education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clinicians (Experimental): Clinician participants will all have access to any clinical implementation strategies that are developed and disseminated in the project.
  Interventions: Other: Clinical implementation strategies
- Patients-Survey Cohort (No Intervention): Patient participants will be observationally followed via survey during the study to monitor patient-reported outcomes.
- Patients-Chart Review Only (No Intervention): Patients who are not in the survey study but who meet other eligibility criteria will undergo chart review to provide electronic health record-based outcomes.

INTERVENTIONS:
Other: Clinical implementation strategies — Clinical implementation strategies, selected based on ED clinician survey/interview findings from Aim 1 using the Implementing Promoting Action on Research Implementation in Health Services (i-PARIHS) implementation science framework
  Arms: Clinicians

SUMMARY:
The purpose of this study is to develop and validate ways to provide better patient education and clinical management for individuals who go to the emergency department (ED) with concussion or mild traumatic brain injury (mTBI).

DETAILED DESCRIPTION:
The study will address three aims: (1) identify factors that help and hinder providing in-ED education to patients with mTBI prior to discharge; (2) examine the impact of tailored implementation strategies on ED providers' provision of in-ED patient education; and (3) evaluate the impact of providing patient education in the ED and through a mobile Health (mHealth) tool post-discharge on patient-level outcomes after mTBI.

ELIGIBILITY:
Inclusion Criteria:

ED clinicians:

• Faculty attending physician, advanced practice professional (APP), resident, fellow, or nurse who practices in an eligible Froedtert & Medical College of Wisconsin (MCW) emergency department

Patients-Survey Cohort:

* Seen and discharged from a Froedtert & MCW emergency department.
* Age 18 or older.
* Has a clinical diagnosis of TBI, as reflected by a relevant International Classification of Disease-10th Edition (ICD-10) code or other evidence (e.g., diagnosis and educational information in the After Visit Summary)
* Speaks English or Spanish.

Patients-Chart Review Only:

* Seen and discharged from a Froedtert & MCW emergency department.
* Age 18 or older.
* Has a clinical diagnosis of TBI, as reflected by a relevant ICD-10 code or other evidence (e.g., diagnosis and educational information in the After Visit Summary).

Exclusion Criteria:

ED clinicians:

• Providers that do not practice in a Froedtert & Medical College of Wisconsin emergency department.

Patients-Survey Cohort.

* In protective custody.
* On psychiatric hold.
* Is not own decision maker (e.g., activated healthcare power of attorney).
* Indicated Do Not Contact in their research contact preferences.
* Left the emergency department prematurely (e.g., against medical advice).
* History of serious health condition that, in the opinion of the investigator, would interfere with engagement in or validity of the survey (e.g., active thought disorder; terminal cancer; dementia).

Patients-Chart Review Only:

• Minors under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5831 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in patient-level penetration-electronic health record (EHR) | Pre-intervention baseline period (estimated study onset to 1 year later); post- intervention follow-up period (estimated 18 months from study onset to 1 year later)
  Change in the percentage of concussion/mTBI-related encounters for which an mTBI patient handout was documented in the Epic After Visit Summary (Aim 2 outcome)
Change in patient-level penetration-patient reported outcome (PRO) | Pre-intervention baseline period (estimated study onset to 1 year later); post- intervention follow-up period (estimated 18 months from study onset to 1 year later)
  Change in the percentage of concussion/mTBI-related encounters for which patients reported having received mTBI patient education before ED discharge (Aim 2 outcome)
Self-efficacy to manage mTBI symptoms | Day 1 post-ED visit, Day 30 post-ED visit
  Patient ratings on the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Self-Efficacy for Managing Symptoms, a 20-point scale based on 4 Likert-type items with 5 response options each (higher scores = more confidence) (Aim 3 outcome).
mTBI symptom burden | Day 1 post-ED visit, Day 30 post-ED visit
  Patient-rated Rivermead Post Concussion Symptoms Questionnaire total score (range 0-64; higher scores = more severe injury-related symptoms) (Aim 3 outcome).

SECONDARY OUTCOMES:
Change in percentage of trauma cases resulting in mTBI diagnosis | Pre-intervention baseline period (estimated study onset to 1 year later); post-intervention follow-up period (estimated 18 months from study onset to 1 year later)
  Change in the percentage of ED encounters for a traumatic injury resulting in a diagnosis of concussion or mTBI
Patient-rated mTBI knowledge | Day 30 post-ED visit
  Patient-rated mTBI knowledge, measured with a 24-item True/False scale (total score range 0-24; higher scores = greater knowledge). Questions ask about common and uncommon mTBI symptoms and common misconceptions about mTBI signs and recovery.
Patient-rated clinical care satisfaction at Day 1 | Day 1 post-ED visit
  Collected on a 5-point scale with the options Very Satisfied, Somewhat Satisfied, Neither Satisfied Nor Dissatisfied, Somewhat Dissatisfied, and Very Dissatisfied. The question is "How satisfied are you with the care you received for head injury in the Emergency Department?"
Patient-rated clinical care satisfaction at Day 30 | Day 30 post-ED visit
  Collected on a 5-point scale with the options Very Satisfied, Somewhat Satisfied, Neither Satisfied Nor Dissatisfied, Somewhat Dissatisfied, and Very Dissatisfied. The question is "How satisfied are you with the care you received for head injury since leaving the emergency department?"

OTHER OUTCOMES:
Change in clinician ratings to the Acceptability of Intervention Measure | Pre-intervention survey period (study onset through roughly 6 months later); post- intervention survey period (roughly 18 months from study onset to 6 months later)
  ED clinician responses to the Acceptability of Intervention Measure (AIM), a 4 item scale with 5-point Likert-type items scaled from 1 (completely disagree) to 5 (completely agree). Total scores reflect the mean item rating (range 1 to 5); higher scores reflect greater acceptability. (Aim 2 outcome; Aim 1 will characterize pre-implementation baseline data only)
Change in clinician ratings to the Intervention Appropriateness Measure | Pre-intervention survey period (study onset through roughly 6 months later); post- intervention survey period (roughly 18 months from study onset to 6 months later)
  ED clinician responses to the Intervention Appropriateness Measure (IAM), a 4 item scale with 5-point Likert-type items scaled from 1 (completely disagree) to 5 (completely agree). Total scores reflect the mean item rating (range 1 to 5); higher scores reflect greater appropriateness. (Aim 2 outcome; Aim 1 will characterize pre-implementation baseline data only)
Change in clinician ratings to the Feasibility of Intervention Measure | Pre-intervention survey period (study onset through roughly 6 months later); post- intervention survey period (roughly 18 months from study onset to 6 months later)
  ED clinician responses to the Feasibility of Intervention Measure (FIM), a 4 item scale with 5-point Likert-type items scaled from 1 (completely disagree) to 5 (completely agree). Total scores reflect the mean item rating (range 1 to 5); higher scores reflect greater feasibility. (Aim 2 outcome; Aim 1 will characterize pre-implementation baseline data only)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified raw data for the Patient-Survey Cohort will be made available on the Open Data Commons for Traumatic Brain Injury (ODC-TBI)

REFERENCES:
- [Background] King NS, Crawford S, Wenden FJ, Moss NE, Wade DT. The Rivermead Post Concussion Symptoms Questionnaire: a measure of symptoms commonly experienced after head injury and its reliability. J Neurol. 1995 Sep;242(9):587-92. doi: 10.1007/BF00868811. PMID 8551320
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459